CLINICAL TRIAL: NCT02243826
Title: Impact of 50% Nitrous Oxide Inhalation on Pain and Anxiety Induced by Lumbar Puncture: a Double-blind Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-206; 2014-001452-28
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Lumbar Puncture
Keywords: Lumbar puncture; Adults; Nitrous oxide; Procedural pain; Procedural anxiety
MeSH Terms: conditions — Pain, Procedural | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- N20 (Experimental): One group will inhale N2O for the 5 minutes before the puncture and during the rest of the procedure.
  Interventions: Drug: 50:50 mixture of nitrous oxide/oxygen
- compressed air (Other): The second group will inhale compressed air during the same period of time
  Interventions: Drug: 50:50 mixture of nitrous oxide/oxygen

INTERVENTIONS:
Drug: 50:50 mixture of nitrous oxide/oxygen

SUMMARY:
This study is designed to evaluate the analgesic effect of nitrous oxide (N2O) on the pain induced during lumbar puncture.

DETAILED DESCRIPTION:
Nitrous oxide (N2O) has analgesic and anxiolytic properties that are known for more than a century. Nonetheless, it's use during lumbar puncture in adults has never been investigated properly.

Thus, this study is designed to evaluate the analgesic effect of N2O on the pain induced during lumbar puncture.

Patients with scheduled lumbar puncture realized for diagnosis purposes will be randomized in 2 groups. One group will inhale N2O for the 5 minutes before the puncture and during the rest of the procedure. The second group will inhale compressed air during the same period of time. Neither the investigator realizing the lumbar puncture, nor the patient will know which type of gaz they are inhaling (double-blinding).

The maximal pain level that occurred during the procedure will be evaluated on a Numerical Rating Scale (NRS). NRS will also be used to evaluate the maximal anxiety induced by the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming in the neurology department for a scheduled lumbar puncture
* 18 to 60 years.
* no previous use of nitrous oxide

Exclusion Criteria:

* contra-indication to nitrous oxide use
* Body Mass Index>35
* Mini Mental State Examination <26/30
* Temperature >38°C
* Confusion
* Patient unable to communicate verbaly

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Maximal pain level during the procedure | at day 1

SECONDARY OUTCOMES:
Maximal anxiety level during the procedure | at day 1
Anxiety evaluated by 2 questionnaires: the Hospital Anxiety and Depression (HAD) State Trait Anxiety Inventory (STAI) | at day 1
Proportion of patients presenting side effects | at day 1
Total duration of the lumbar puncture | at day 1
Proportion of patients that would accept another lumbar puncture in the same conditions | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CLAVELOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France